CLINICAL TRIAL: NCT02043678
Title: A Phase III Randomized, Double-blind, Placebo-controlled Trial of Radium-223 Dichloride in Combination With Abiraterone Acetate and Prednisone/Prednisolone in the Treatment of Asymptomatic or Mildly Symptomatic Chemotherapy-naïve Subjects With Bone Predominant Metastatic Castration-resistant Prostate Cancer(CRPC)
Brief Title: Radium-223 Dichloride and Abiraterone Acetate Compared to Placebo and Abiraterone Acetate for Men With Cancer of the Prostate When Medical or Surgical Castration Does Not Work and When the Cancer Has Spread to the Bone, Has Not Been Treated With Chemotherapy and is Causing no or Only Mild Symptoms
Acronym: ERA 223
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15396; 2013-003438-33 (EudraCT Number)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms
Keywords: Phase III; Radium-223 dichloride; Abiraterone acetate; Combination therapy; Chemotherapy-naive; Bone metastasis; Castration-resistant prostate cancer (CRPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Saline Solution; abiraterone; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Radium-223 dichloride + Abi/Pred (Experimental): Participants received 6 intravenous (IV) administrations of radium-223 dichloride 50 kiloBecquerel per kilogram (kBq/kg) (55 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update) body weight at intervals of 4 weeks, along with oral abiraterone acetate tablets 1000 milligrams (mg) every day plus prednisone/prednisolone 5 mg twice daily (abi/pred) for 6 cycles, followed by abi/pred until an on-study symptomatic skeletal event (SSE) occurred (or other withdrawal criteria were met)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Abiraterone; Drug: Prednisone/Prednisolone
- Placebo + Abi/Pred (Placebo Comparator): Participants received 6 IV administrations of placebo matched to radium-223 dichloride at intervals of 4 weeks, along with abi/pred for 6 cycles, followed by abi/pred until an on-study SSE occurred (or other withdrawal criteria were met)
  Interventions: Drug: Matching placebo (normal saline); Drug: Abiraterone; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — 50 kiloBecquerel per kilogram (kBq/kg) (55 kBq/kg after implementation of NIST update) body weight, intravenous injection (IV-slow bolus), every 4 weeks for 6 cycles
  Arms: Radium-223 dichloride + Abi/Pred
Drug: Matching placebo (normal saline) — Intravenous injection ( IV-slow bolus), every 4 weeks for 6 cycles
  Arms: Placebo + Abi/Pred
Drug: Abiraterone — 1000 mg once daily, oral, with best supportive care
Drug: Prednisone/Prednisolone — 5 mg twice daily, oral, with best supportive care

SUMMARY:
To determine if the addition of radium-223 dichloride to standard treatment is able to prolong life and to delay events specific for prostate cancer which has spread to the bone, such as painful fractures or bone pain which needs to be treated with an X-ray machine.

DETAILED DESCRIPTION:
This study is a phase III multinational, multicenter,randomized, double blind, placebo controlled, study with a randomization allocation ratio of 1:1 (radium-223 dichloride plus abiraterone acetate plus prednisone/prednisolone: placebo plus abiraterone acetate plus prednisone/prednisolone). Until the final overall survival (OS) analysis, the study period consisted of screening / randomization, treatment, active follow-up with clinic visits, active follow-up without clinic visits, and longterm follow-up phases. Up until this point, subjects received study treatment (radium-223 dichloride or placebo in addition to abiraterone acetate plus prednisone / prednisolone for the first 6 cycles followed by abiraterone acetate plus prednisone / prednisolone thereafter) until an on-study SSE occurred (or other withdrawal criteria were met). After the final OS analysis (after implementation of Amendment 7), in order to reduce the burden to study subjects, evaluation of efficacy and exploratory endpoints will be discontinued, except for symptomatic skeletal event (SSE) and OS. Subjects who are discontinued from study treatment will initiate the long-term follow-up period; therefore, active follow-up periods will no longer be applicable. Subjects who are in active follow-up at the time of Amendment 7 is implemented should have the end of active follow-up completed (protocol driven decision) and should be directly transitioned into the extended safety follow-up study. Long term follow-up will continue until the subject dies, is lost to follow-up, withdraws informed consent, actively objects to collection of further data , or is transitioned to the extended safety follow-up study. Subjects will be followed for safety for up to 7 years, which eventually will be completed in this study or in the extended safety follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Male subjects of age ≥ 18 years
* Prostate cancer progression documented by prostate specific antigen (PSA) according to the Prostate Cancer Working Group 2 (PCWG2) criteria or radiological progression according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
* Two or more bone metastases on bone scan within 4 weeks prior to randomization with no lung, liver, other visceral and/or brain metastasis
* Asymptomatic or mildly symptomatic prostate cancer
* Subjects who received combined androgen blockade with an anti-androgen must have shown PSA progression after discontinuing the anti-androgen prior to enrollment
* Maintenance of medical castration or surgical castration with testosterone less than 50 ng/dL (1.7nmol/L)
* Eastern Cooperative Oncology Group performance status (ECOG PS) score 0 or 1

Exclusion Criteria:

* Prior cytotoxic chemotherapy for the treatment of CRPC, including taxanes, mitoxantrone and estramustine
* Any chronic medical condition requiring a higher dose of corticosteroid than 5 mg prednisone/prednisolone twice daily
* Pathological finding consistent with small cell carcinoma of the prostate
* History of visceral metastasis, or presence of visceral metastasis detected by screening imaging examinations
* History of or known brain metastasis
* Malignant lymphadenopathy exceeding 3 cm in short-axis diameter
* Blood transfusion or erythropoietin stimulating agents prior 4 weeks of screening and during the whole screening period before randomization
* Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Subjects with history of spinal cord compression should have completely recovered
* Use of opiate analgesics for cancer-related pain, including codeine and dextropropoxyphene, currently or anytime during the 4- week period prior to randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2014-03-30 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (150):
- United States (28):
  - Anchorage, Alaska
  - Tucson, Arizona
  - Oceanside, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - Atlanta, Georgia
  - Jeffersonville, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Traverse City, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Poughkeepsie, New York
  - Syracuse, New York
  - Bala-Cynwyd, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Norfolk, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Wheeling, West Virginia
- Australia (8):
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Adelaide, South Australia
  - East Bentleigh, Victoria
  - Fitzroy, Victoria
  - Heidelberg, Victoria
  - East Melbourne
  - Randwick
- Belgium (4):
  - Brussels
  - Bruxelles - Brussel
  - Edegem
  - Ghent
- Brazil (5):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Barretos/SP, São Paulo
  - São Paulo, São Paulo
  - São Paulo
- Canada (8):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Finland (4):
  - Helsinki
  - Kuopio
  - Seinäjoki
  - Tampere
- France (6):
  - Besançon
  - Bordeaux
  - Paris
  - Poitiers
  - Saint-Herblain
  - Toulouse
- Germany (7):
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Marburg, Hesse
  - Münster, North Rhine-Westphalia
  - Dresden, Saxony
  - Jena, Thuringia
  - Berlin
- Israel (9):
  - Afula
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Italy (7):
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Cagliari, Sardinia
  - Trento, Trentino-Alto Adige
  - Cortona, Tuscany
- Japan (27):
  - Nagoya, Aichi-ken
  - Hirosaki, Aomori
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Tsukuba, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Kita-gun, Kagawa-ken
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Sayama, Osaka
  - Hamamatsu, Shizuoka
  - Bunkyo-Ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Koto-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Ube, Yamaguchi
  - Chiba
  - Fukuoka
  - Kumamoto
  - Miyazaki
  - Nagasaki
- Netherlands (3):
  - Amsterdam
  - Nijmegen
  - Zwolle
- Norway (3):
  - Bodø
  - Lørenskog
  - Oslo
- Poland (4):
  - Gdansk
  - Gdynia
  - Gliwice
  - Poznan
- Russia (2):
  - Moscow
  - Obninsk
- Singapore, Singapore
- Spain (8):
  - Badalona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Málaga, Málaga
  - Oviedo, Principality of Asturias
  - Barcelona
  - Madrid
  - Pamplona
  - Seville
- Sweden (5):
  - Linköping
  - Stockholm
  - Sundsvall
  - Umeå
  - Vaxjo
- United Kingdom (11):
  - Edinburgh, Lothian
  - Bebington, Merseyside
  - Northwood, Middlesex
  - Guildford, Surrey
  - Sutton, Surrey
  - Newcastle upon Tyne, Tyne and Wear
  - Coventry, West Midlands
  - Belfast
  - Leeds
  - London
  - Romford

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Result] Smith M, Parker C, Saad F, Miller K, Tombal B, Ng QS, Boegemann M, Matveev V, Piulats JM, Zucca LE, Karyakin O, Kimura G, Matsubara N, Nahas WC, Nole F, Rosenbaum E, Heidenreich A, Kakehi Y, Zhang A, Krissel H, Teufel M, Shen J, Wagner V, Higano C. Addition of radium-223 to abiraterone acetate and prednisone or prednisolone in patients with castration-resistant prostate cancer and bone metastases (ERA 223): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):408-419. doi: 10.1016/S1470-2045(18)30860-X. Epub 2019 Feb 6. PMID 30738780
- [Derived] Shore N, Higano CS, George DJ, Sternberg CN, Saad F, Tombal B, Miller K, Kalinovsky J, Jiao X, Tangirala K, Sartor O. Concurrent or layered treatment with radium-223 and enzalutamide or abiraterone/prednisone: real-world clinical outcomes in patients with metastatic castration-resistant prostate cancer. Prostate Cancer Prostatic Dis. 2020 Dec;23(4):680-688. doi: 10.1038/s41391-020-0236-0. Epub 2020 May 13. PMID 32404868
- [Derived] Matsubara N, Kimura G, Uemura H, Uemura H, Nakamura M, Nagamori S, Mizokami A, Kikukawa H, Hosono M, Kinuya S, Krissel H, Siegel J, Kakehi Y. A randomized, double-blind, comparison of radium-223 and placebo, in combination with abiraterone acetate and prednisolone, in castration-resistant metastatic prostate cancer: subgroup analysis of Japanese patients in the ERA 223 study. Int J Clin Oncol. 2020 Apr;25(4):720-731. doi: 10.1007/s10147-019-01589-6. Epub 2019 Dec 10. PMID 31823152
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 19 countries between 30 March 2014 (first participant first visit) and 08 February 2024 (last participant last visit).
Pre-assignment Details: Overall, 1144 participants were screened. Of them, 338 participants did not complete screening, 806 participants were randomized to treatment and 786 participants received study treatment. 2 participants randomized to the placebo treatment group unintentionally received 1 radium-223 dichloride dose during the treatment period.
Period: Overall Study
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Started | 401 | 405
Treated | 390 | 396
Completed (Completed treatment) | 0 | 0
Not Completed | 401 | 405
Not completed — Never treated | 11 | 9
Not completed — AE with clinical progressive disease(PD) | 20 | 19
Not completed — AE without clinical PD | 54 | 36
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 10 | 14
Not completed — Clinical PD | 114 | 148
Not completed — Radiological PD | 100 | 90
Not completed — Protocol-driven decision point | 59 | 58
Not completed — Withdrawal by Subject | 16 | 20
Not completed — Protocol Violation | 1 | 0
Not completed — Deterioration of general conditions | 1 | 1
Not completed — Logistical difficulties | 2 | 0
Not completed — Non-compliance with study drug | 3 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Subject decision | 0 | 1
Not completed — Switching to other therapy | 3 | 2
Not completed — Ongoing with commercial abiraterone/prednisone outside study | 1 | 1
Not completed — Missing | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set (ITT) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred | Total
Number analyzed (Participants) | 401 | 405 | 806
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (8.5) | 71.4 (8.4) | 71.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 401 | 405 | 806
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 23 | 40
  Not Hispanic or Latino | 361 | 355 | 716
  Unknown or Not Reported | 23 | 27 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 79 | 78 | 157
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 285 | 284 | 569
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 26 | 52
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: ITT analysis set with evaluable number of participants
  Kilograms (kg)
    number analyzed (Participants) | 396 | 400 | 796
    (all) | 82.19 (16.75) | 82.40 (16.01) | 82.30 (16.37)
Stage of prostate cancer at diagnosis (Tumor Node Metastasis [TNM] Classification) [Count of Participants; unit: Participants] — TNM staging system stands for Tumour, Node, Metastasis. Stage I: cancer is in half of one side of the prostate or less. Stage II: cancer is in more than half of one side of the prostate, completely contained within the prostate gland. Stage III: cancer has broken through the capsule of the prostate gland, and may have spread into tubes that carry semen. Stage IV: cancer has spread into nearby body organs, such as the back passage or bladder; or has spread to nearby lymph nodes; or has spread to other parts of the body outside the pelvis, such as the lungs or liver.
  Participants
    Missing | 19 | 24 | 43
    Stage I | 27 | 18 | 45
    Stage IIA | 22 | 20 | 42
    Stage IIB | 34 | 49 | 83
    Stage III | 102 | 88 | 190
    Stage IV | 197 | 206 | 403
Cancer pain assessment by Brief Pain Inventory-Short Form (BPI-SF) [Count of Participants; unit: Participants] — The BPI-SF is a short, self-administered questionnaire with 11 items designed to evaluate the intensity of, and the impairment caused by pain. Four items measure pain intensity (pain now, average pain, worst pain, and least pain) using 0 ("no pain") to 10 ("pain as bad as you can imagine") numeric rating scales, and 7 items measure the level of interference with function caused by pain (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life) using 0 (no interference) to 10 (complete interference) rating scales.
  Participants
    Missing | 25 | 33 | 58
    Asymptomatic (Worst pain score = 0) | 195 | 198 | 393
    Mildly Symptomatic (Worst pain score 1 - 3) | 181 | 174 | 355
Gleason score at diagnosis [Count of Participants; unit: Participants] — The Gleason score is an indication of prognosis based on prostate pathology. The total score ranges from 2 to 10 (ie: "1+1" to "5+5") with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5).
  Participants
    Missing | 15 | 18 | 33
    Less than (<) 8 | 140 | 154 | 294
    Greater than or equal to (>=) 8 | 246 | 233 | 479
Prostate-specific antigen [Mean (Standard Deviation); unit: Micrograms per liter (ug/L)] — Population: ITT set with evaluable number of participants.
  Micrograms per liter (ug/L)
    number analyzed (Participants) | 396 | 401 | 797
    (all) | 92.39 (191.62) | 92.33 (328.00) | 92.36 (268.85)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern cooperative oncology group (ECOG) performance status: 0= Fully active, able to carry on all pre-disease performance without restriction; 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2= Ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3= Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4= Completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  Participants
    Missing | 2 | 3 | 5
    0 | 262 | 281 | 543
    1 | 137 | 121 | 258
Extent of Disease [Count of Participants; unit: Participants]
  Normal or abnormal because of benign bone disease | 2 | 0 | 2
  < 6 metastases | 134 | 141 | 275
  6-20 metastases | 175 | 181 | 356
  >20 lesions but not a superscan | 71 | 70 | 141
  Superscan | 19 | 13 | 32

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Skeletal Event Free Survival (SSE-FS)
Description: SSE-FS was defined as time (months) from randomization to the earliest of onset date of skeletal symptoms treated with external beam radiotherapy (EBRT), onset date of pathological bone fracture, onset date of spinal cord compression, procedure date of tumor-related orthopedic surgery, or death from any cause. Participants who died without prior SSE and ≥ 13 weeks after the last SSE assessment are censored at the last SSE assessment date. Participants alive at the survival cut-off date are censored at the last date known to be alive. Participants with multiple events are only counted for the category in which the first event occurred. If multiple SSE (component events) occur on the same date for 1 participant, the participant is only counted into 1 category in the order of: spinal cord compression > bone fracture > orthopedic surgery > EBRT.
Time Frame: From randomization until first onset of on-study symptomatic skeletal event (SSE) or death, up to 47 months
Population: Intent-to-Treat (ITT) analysis set (included all randomized participants)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 401 | 405
Months | 22.3 [20.4 to 24.8] | 26.0 [21.8 to 28.3]
Statistical Analysis 1: Comparison: Radium-223 Dichloride + Abi/Pred vs Placebo + Abi/Pred; Test type: Superiority; p = 0.2636, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.122, 95% CI 2-sided [0.917 to 1.374]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (months) from the date of randomization to the date of death due to any cause. Participants alive at the survival cut-off date were censored at the last date known to be alive.
Time Frame: From randomization until death from any cause, up to 67 months
Population: ITT analysis set (included all randomized participants)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 401 | 405
Months | 30.1 [27.5 to 33.2] | 34.8 [31.5 to 37.6]
Statistical Analysis 1: Comparison: Radium-223 Dichloride + Abi/Pred vs Placebo + Abi/Pred; Test type: Superiority; p = 0.1194, Cox Proportional Hazards model; Hazard Ratio (HR) = 1.151, 95% CI 2-sided [0.964 to 1.374]

3. Secondary Outcome: Radiological Progression Free Survival (rPFS)
Description: rPFS was defined as the time (months) from the date of randomization to the date of confirmed radiological progression or death (if death occurred before progression) based on independent assessment.
Time Frame: From randomization until the date of confirmed radiological progression or death, up to 47 months
Population: ITT analysis set (included all randomized participants)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 401 | 405
Months | 11.2 [9.1 to 11.8] | 12.4 [10.8 to 14.5]
Statistical Analysis 1: Comparison: Radium-223 Dichloride + Abi/Pred vs Placebo + Abi/Pred; Test type: Superiority; p = 0.1283, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.152, 95% CI 2-sided [0.960 to 1.383]

4. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the interval from randomization to the first date a participant experienced pain progression assessed by Brief Pain Inventory-Short Form and defined as: an increase of 2 or more points in the average worst pain score (WPS) from baseline observed at 2 consecutive evaluations ≥4 weeks apart or initiation of short- or long-acting opioid use for pain for participants with WPS 0 at baseline; an increase of 2 or more points in the average WPS from baseline observed at 2 consecutive evaluations ≥4 weeks apart and an average WPS of ≥4 OR initiation of short- or long-acting opioid use for pain for participants with WPS 1 to 3 at baseline. Participants without pain progression at end of study are censored at the last date known to have not progressed: last evaluation date for pain scores or last visit when recorded opiate use, whichever is last. Participants with no on-study assessment or no baseline assessment are censored at the date of randomization.
Time Frame: From randomization until the date of pain progression based on pain score, up to 47 months
Population: ITT analysis set (included all randomized participants)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 401 | 405
Months | 14.4 [11.1 to 20.1] | 18.7 [15.4 to 23.1]
Statistical Analysis 1: Comparison: Radium-223 Dichloride + Abi/Pred vs Placebo + Abi/Pred; Test type: Superiority; p = 0.1669, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.145, 95% CI 2-sided [0.945 to 1.389]

5. Secondary Outcome: Time to Cytotoxic Chemotherapy
Description: Time to cytotoxic chemotherapy is time (months) from randomization to the earliest date of the first cytotoxic chemotherapy. Participants who have not started cytotoxic chemotherapy during the study were censored at the last assessment date.
Time Frame: From randomization until the date of first cytotoxic chemotherapy, up to 47 months
Population: ITT analysis set (included all randomized participants)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 401 | 405
Months | 29.5 [26.5 to 35.7] | 28.5 [23.7 to NA] — Upper limit cannot be estimated due to censored data.
Statistical Analysis 1: Comparison: Radium-223 Dichloride + Abi/Pred vs Placebo + Abi/Pred; Test type: Superiority; p = 0.7871, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.033, 95% CI 2-sided [0.816 to 1.308]

6. Secondary Outcome: Time to Opiate Use for Cancer Pain
Description: Time to opiate use for cancer pain was defined as the interval from the date of randomization to the date of opiate use.
Time Frame: From randomization until the date of opiate use, up to 47 months
Population: ITT analysis set excluding participants who had opiate use at baseline
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 398 | 392
Months | 19.0 [14.4 to 23.2] | 22.6 [18.0 to 25.7]
Statistical Analysis 1: Comparison: Radium-223 Dichloride + Abi/Pred vs Placebo + Abi/Pred; Test type: Superiority; p = 0.2467, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.126, 95% CI 2-sided [0.921 to 1.378]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant in the study. A serious adverse event (SAE) was any untoward medical occurrence that at any dose was resulting in death, was life-threatening, requires hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity. A treatment-emergent AEs (TEAEs) or serious TEAEs was defined as any event that started on or after the first dose of the study treatment and during the treatment period and was not a continuation of a pretreatment event or started before the first dose and worsened after the first dose or the treatment period. Drug-related TEAEs or serious TEAEs were those with "reasonable causal relationship" to the study treatment decided by the investigators.
Time Frame: From start of study treatment until the end of the treatment period, up to 110 months
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants
  Any TEAE | 382 | 387
  Any drug-related TEAE | 265 | 273
  Radium-223/Placebo-related TEAE | 92 | 91
  Any serious TEAE | 178 | 178
  Any drug-related serious TEAE | 32 | 30
  Radium-223/Placebo-related serious TEAE | 12 | 7

8. Secondary Outcome: Number of Participants With Radium-223/Placebo-related Treatment-emergent Adverse Events Per Maximum Intensity
Description: An adverse event (AE) was any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant in the study. A serious adverse event (SAE) was any untoward medical occurrence that at any dose was resulting in death, was lifethreatening, requires hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity. A treatment-emergent AEs (TEAEs) or serious TEAEs was defined as any event that started on or after the first dose of the study treatment and during the treatment period and was not a continuation of a pretreatment event or started before the first dose and worsened after the first dose or the treatment period. Radium-223/placebo-related TEAEs or serious TEAEs were those with "reasonable causal relationship" to radium-223 or placebo decided by the investigators.
Time Frame: From start of study treatment until the end of the treatment period, up to 110 months
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants
  TEAE - Grade 1 | 43 | 53
  TEAE - Grade 2 | 28 | 23
  TEAE - Grade 3 | 20 | 13
  TEAE - Grade 4 | 1 | 2
  Serious TEAE - Grade 2 | 3 | 0
  Serious TEAE - Grade 3 | 9 | 5
  Serious TEAE - Grade 4 | 0 | 2

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Additional Primary Malignancies
Description: Treatment-emergent additional primary malignancies were adverse events identified as additional primary malignancies that occurred after start of study treatment until the end of the treatment period.
Time Frame: From start of study treatment until the end of the treatment period, up to 110 months
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants | 32 | 30

10. Secondary Outcome: Number of Participants With Treatment-emergent Bone Fractures
Description: Treatment-emergent fractures were adverse events identified as fractures that occurred after start of study treatment until the end of the treatment period. All bone fractures and bone-associated events (e.g., osteoporosis) were reported as either AEs, or SAEs if the criteria of SAE were met, regardless of the investigator's causality assessment.
Time Frame: From start of study treatment until the end of the treatment period, up to 110 months
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants | 110 | 51

11. Secondary Outcome: Number of Participants With Post-treatment Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant in the study. Any bleeding event occurring during the study was not documented as an AE because this event was planned to be captured in the assessment of efficacy. AEs that started after the treatment period were defined as post-treatment AEs. Drug-related AEs were those with "reasonable causal relationship" to the study treatment decided by the investigators.
Time Frame: After the treatment period, up to 48.5 months in active follow-up and 74.9 months in long-term follow-up
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants
  Any events | 148 | 138
  Any drug-related events | 20 | 10
  Any chemotherapy-related events | 31 | 34

12. Secondary Outcome: Number of Participants With Any Study Drug-related Post-treatment Adverse Events Per Maximum Intensity
Description: as for outcome 11
Time Frame: After the treatment period, up to 48.5 months in active follow-up and 74.9 months in long-term follow-up
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants
  Grade 1 | 34 | 4
  Grade 2 | 9 | 3
  Grade 3 | 6 | 3
  Grade 4 | 1 | 0

13. Secondary Outcome: Number of Participants With Post-treatment Additional Primary Malignancies
Description: Post-treatment additional primary malignancies were adverse events identified as additional primary malignancies that started after the treatment period.
Time Frame: After the treatment period, up to 48.5 months in active follow-up and 74.9 months in long-term follow-up
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants | 7 | 7

14. Secondary Outcome: Number of Participants With Post-treatment Chemotherapy-related Blood and Lymphatic System Disorders
Description: Post-treatment blood and lymphatic system disorders were adverse events identified as blood and lymphatic system disorders that occurred after the end of the treatment period until participant died, was lost to follow-up, withdrew informed consent, actively objected to collection of further data, or was transitioned to the extended safety follow-up study.
Time Frame: After the treatment period, up to 48.5 months in active follow-up and 74.9 months in long-term follow-up
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants
  Anaemia | 5 | 4
  Myelosuppression | 1 | 0
  Febrile neutropenia | 5 | 8
  Leukopenia | 1 | 0
  Neutropenia | 8 | 3
  Pancytopenia | 0 | 1
  Thrombocytopenia | 2 | 2

15. Secondary Outcome: Number of Participants With Post-treatment Bone Fractures
Description: Post-treatment fractures were adverse events identified as fractures that occured after the end of the treatment period until participant died, was lost to follow-up, withdrew informed consent, actively objected to collection of further data, or was transitioned to the extended safety follow-up study. All bone fractures and bone-associated events (e.g., osteoporosis), were reported as either AEs, or SAEs if the criteria of SAE were met, regardless of the investigator's causality assessment.
Time Frame: After the treatment period, up to 48.5 months in active follow-up and 74.9 months in long-term follow-up
Population: Safety analysis set (SAF): included all randomized participants who received at least one dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
Number analyzed (Participants) | 392 | 394
Participants
  Ankle fracture | 0 | 1
  Craniofacial fracture | 1 | 0
  Femur fracture | 1 | 0
  Fibula fracture | 0 | 1
  Foot fracture | 1 | 0
  Jaw fracture | 1 | 0
  Patella fracture | 1 | 0
  Radius fracture | 1 | 0
  Rib fracture | 0 | 1
  Spinal compression fracture | 0 | 2
  Thoracic vertebral fracture | 0 | 1
  Traumatic fracture | 0 | 1
  Osteoporotic fracture | 6 | 0
  Pathological fracture | 14 | 14

ADVERSE EVENTS:
Time Frame: From start of study treatment until last contact, up to 110 months in treatment period, 48.5 months in active follow-up and 74.9 months in long-term follow-up.
Description: Adverse events (AEs) included any event arising or worsening from the start of the study treatment. All occurrences of additional malignancies, chemotherapy-related events, bone fractures and bone associated events were reported as AE regardless of the investigator's causality assessment.
Arm/Group | Radium-223 Dichloride + Abi/Pred | Placebo + Abi/Pred
All-Cause Mortality (participants affected / at risk) | 287/392 | 290/394
Serious Adverse Events (participants affected / at risk) | 193/392 | 191/394
Other Adverse Events (participants affected / at risk) | 368/392 | 376/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 Dichloride + Abi/Pred (N=392) | Placebo + Abi/Pred (N=394)
Anaemia (Blood and lymphatic system disorders) | 9 (19) | 4 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (8) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (5) | 4 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 8 (9)
Atrial flutter (Cardiac disorders) | 1 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (3) | 3 (6)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (4) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (2) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Inborn error of metabolism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Primary adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (2)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (4)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Overflow diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (2) | 4 (6)
Condition aggravated (General disorders) | 2 (3) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Sudden death (General disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 9 (13) | 13 (19)
Physical deconditioning (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 12 (15) | 16 (20)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (4) | 4 (7)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (6)
Urinary tract infection (Infections and infestations) | 18 (21) | 11 (13)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Wound infection (Infections and infestations) | 1 (3) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 6 (12)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Acute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (4) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (2)
Arthritis infective (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Neurocryptococcosis (Infections and infestations) | 1 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (6) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudophakic bullous keratopathy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (6) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (3)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (11)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 11 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (8)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 9 (14) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 10 (15) | 4 (4)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Jaw fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (1)
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (8) | 6 (13)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (6)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (3)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 8 (24)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Alexia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (3) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Spinal cord compression (Nervous system disorders) | 7 (7) | 9 (9)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (3) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (6) | 4 (5)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (5) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (3) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (7)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (3)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (3)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (5) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (4) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 Dichloride + Abi/Pred (N=392) | Placebo + Abi/Pred (N=394)
Anaemia (Blood and lymphatic system disorders) | 64 (135) | 62 (129)
Abdominal pain (Gastrointestinal disorders) | 23 (24) | 17 (20)
Constipation (Gastrointestinal disorders) | 71 (84) | 83 (102)
Diarrhoea (Gastrointestinal disorders) | 71 (111) | 71 (102)
Dyspepsia (Gastrointestinal disorders) | 20 (23) | 16 (17)
Nausea (Gastrointestinal disorders) | 76 (92) | 69 (77)
Vomiting (Gastrointestinal disorders) | 41 (49) | 42 (48)
Asthenia (General disorders) | 39 (50) | 44 (61)
Chest pain (General disorders) | 20 (22) | 19 (25)
Fatigue (General disorders) | 106 (152) | 97 (140)
Influenza like illness (General disorders) | 15 (19) | 20 (24)
Oedema peripheral (General disorders) | 61 (83) | 68 (81)
Pyrexia (General disorders) | 30 (35) | 34 (50)
Influenza (Infections and infestations) | 22 (23) | 14 (22)
Nasopharyngitis (Infections and infestations) | 31 (40) | 39 (54)
Upper respiratory tract infection (Infections and infestations) | 29 (42) | 35 (47)
Urinary tract infection (Infections and infestations) | 40 (55) | 34 (41)
Fall (Injury, poisoning and procedural complications) | 61 (93) | 52 (78)
Rib fracture (Injury, poisoning and procedural complications) | 22 (37) | 17 (39)
Contusion (Injury, poisoning and procedural complications) | 28 (38) | 33 (41)
Alanine aminotransferase increased (Investigations) | 69 (180) | 61 (151)
Aspartate aminotransferase increased (Investigations) | 61 (127) | 55 (106)
Weight decreased (Investigations) | 23 (37) | 25 (39)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (18) | 23 (50)
Hypokalaemia (Metabolism and nutrition disorders) | 43 (81) | 45 (87)
Decreased appetite (Metabolism and nutrition disorders) | 68 (86) | 54 (58)
Arthralgia (Musculoskeletal and connective tissue disorders) | 106 (170) | 104 (197)
Back pain (Musculoskeletal and connective tissue disorders) | 154 (258) | 140 (214)
Bone pain (Musculoskeletal and connective tissue disorders) | 72 (103) | 76 (101)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 (34) | 30 (34)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 26 (40) | 37 (51)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (20) | 22 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (29) | 24 (27)
Neck pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 26 (32)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 27 (28) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 26 (75) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 53 (75) | 59 (80)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 49 (73) | 28 (43)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 30 (43) | 32 (40)
Spinal pain (Musculoskeletal and connective tissue disorders) | 31 (36) | 27 (34)
Dizziness (Nervous system disorders) | 45 (54) | 37 (44)
Headache (Nervous system disorders) | 31 (46) | 31 (38)
Insomnia (Psychiatric disorders) | 34 (37) | 26 (27)
Haematuria (Renal and urinary disorders) | 32 (45) | 21 (29)
Pelvic pain (Reproductive system and breast disorders) | 12 (16) | 21 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (42) | 42 (53)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 32 (36)
Hypertension (Vascular disorders) | 62 (168) | 83 (221)
Hot flush (Vascular disorders) | 24 (26) | 51 (53)

LIMITATIONS AND CAVEATS:
2 participants randomized to the placebo treatment group unintentionally received 1 radium-223 dichloride dose during the treatment period. These 2 participants are summarized in the radium-223 dichloride treatment group in the safety analysis; while were analyzed as randomized, i.e., in the placebo arm for the efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02043678/Prot_002.pdf
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02043678/SAP_001.pdf